CLINICAL TRIAL: NCT05366218
Title: A Prospective Phase I/II, Single-Arm, Open-Label, Multicentre Study to Evaluate the Safety and Efficacy of Tafasitamab (MOR00208) in Pediatric Patients With Relapsed or Refractory Acute B Lineage Leukemia
Brief Title: Tafasitamab (MOR00208) in Pediatric Patients With Relapsed or Refractory Acute B Lineage Leukemia
Acronym: Anti-CD19-ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-000557-88; 2024-511336-28-00 (EU CTIS Number)
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: ALL, Childhood B-Cell; Acute Lymphoid Leukemia Relapse; Acute Lymphocytic Leukemia Refractory
Keywords: CD19 positive; refractory to standard treatment; relapse
MeSH Terms: conditions — Recurrence | interventions — tafasitamab

STUDY DESIGN:
Intervention Model Description: A Prospective Phase I/II, Single-Arm, Open-Label, Multicentre Study to Evaluate the Safety and Efficacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tafasitamab (Experimental): All patients will receive MOR00208 over 2-3 hours i.v. MOR00208 will be administered on a bi-weekly (every fourteen days) basis with infusions on Days 1 and 15 of each 28-day cycle. Additional doses will be administered on Day 4, Day 8 and Day 22 of Cycle 1 as well as Day 8 and Day 22 of Cycle 2 and Cycle 3.
  Interventions: Biological: Tafasitamab

INTERVENTIONS:
Biological: Tafasitamab — Antibody vaccination
  Other Names: MOR00208

SUMMARY:
The objective of the trial is to evaluate the safety, clinical toxicity and in vivo immunological effects of MOR00208 in pediatric patients with acute lymphoblastic leukemia who showed newly emerging or persistent MRD after a first stem cell transplantation, received stem cell transplantation without having reached a sufficient molecular remission prior to transplant (defined as MRD ≥10E-4) irrespective of MRD after SCT or underwent a second or subsequent stem cell transplantation irrespective of MRD after SCT.

Part I: to determine the recommended dose of MOR00208 in pediatric patients Part II: to evaluate the time until hematological relapse or increase of MRD

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia is the most common malignancy in children. In patients with > 2nd relapse or in patients who relapse after previous stem cell transplantation (SCT), conventional chemotherapy or even subsequent SCT results only in low probabilities for event free survival (1-year EFS ~30%) with a generally poor prognosis. Major cause of death is a subsequent relapse. To date there is no standard therapy available. The aim of this study is to establish an antibody approach as an additional therapy. Therefore, the safety and efficacy of the anti-CD19-antibody tafasitamab in such pediatric very high-risk patients will be evaluated. Patients will be included in the following stages of disease: newly emerging or persistent minimal residual disease (MRD) after a first SCT; SCT without having reached a sufficient molecular remission prior to transplant (defined as MRD ≥10E-4) irrespective of MRD after SCT; underwent a second or subsequent SCT irrespective of MRD after SCT. Tafasitamab will be used as a relapse prophylaxis as well as a treatment for patients with low detectable low MRD. The treatment is intended to reduce the likelihood of overt relapse after SCT in a collective of patients at highest risk of relapse, thereby improving the long-term survival of these patients. The bi-weekly application of anti-CD19-antibody has already shown promising results in compassionate use settings in pediatric patients. Furthermore, the safety of tafasitamab has already been analyzed in multiple studies in adults and has proven to be well tolerable. As a control group published data for these patient groups will be used with a combined 1-year EFS of 30% in which patients have been treated at the current standard of care.

The study consists of 2 parts:

The first part will evaluate safety along with the maximum tolerated dose of tafasitamab in pediatric patients. This will involve intra- and inter-individual dose escalation using pre-determined dose levels before the dose-finding phase is completed. If dose-limiting drug side effects occur during this dose-finding phase, additional patients will be included in the interindividual dose escalation until the maximum tolerated dose of tafasitamab is defined for the remainder of the study. For this dose-finding phase, a minimum of six and a maximum of 25 patients will be included.

Immediately thereafter, the second study phase begins, in which all patients from the dose-finding phase who have not experienced a dose-limiting toxicity, as well as additional enrolled patients, receive the defined maximum tolerated dose of tafasitamab. In this phase of the study, in addition to the continued recording of drug side effects, the efficacy of tafasitamab will be assessed using defined endpoints. A minimum evaluable number of 18 patients is planned for the assessment of these endpoints; to compensate for possible patient dropout during the study, recruitment of a minimum of 20 patients and a maximum of 39 patients, depending on the course of the dose-finding phase, is planned.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 years and < 18 years at enrollment
* B-lineage (CD19 positive) ALL (B, pro-B, pre-B or c-ALL)
* Patients must have either

  * underwent a first allogeneic stem cell transplantation after relapse with one of the following very high-risk somatic molecular alterations:

    * KMT2A::AFF1 [t(4;11) rearrangement
    * TP53 alteration (mutation/deletion)
    * low hypodiploidy (<40 chromosomes, evident or masked)
    * TCF3-PBX1 [t(1;19)]
    * TCF3::HLF [t(17;19)] and irrespective of MRD after SCT or
  * underwent a first allogeneic stem cell transplantation or a CAR T-cell therapy with newly emerging or persistent MRD load posttransplant / post CAR T- cell-treatment or
  * have received stem cell transplantation without having reached a sufficient molecular remission prior to transplant (defined as MRD ≥10E-4) irrespective of MRD after SCT or
  * underwent a second or subsequent allogeneic stem cell transplantation irrespective of MRD after SCT
* Females of childbearing potential (FCBP1) must agree

  * to utilize two reliable forms of contraception simultaneously or practice complete abstinence from heterosexual contact for at least 3 months before starting study drug, while participating in the study (including dose interruptions), and for at least 3 months after study treatment discontinuation and must agree to regular pregnancy testing during this timeframe
  * to abstain from breastfeeding during study participation and 3 months after study drug discontinuation.
* Males must agree

  * to use a latex condom during any sexual contact with FCBP while participating in the study and for 3 months following discontinuation from this study, even if he has undergone a successful vasectomy
  * to refrain from donating semen or sperm during study participation and for 3 months after discontinuation from this study treatment.

Exclusion Criteria:

* Frank relapse (>5% leukemic blasts)
* Philadelphia chromosome-positive (Ph+) ALL
* Ejection fraction <25% on echocardiography
* Cystatin C-clearance <40ml/min
* Liver function abnormalities with bilirubin >4 mg/dL and elevation of transaminases higher than 400 U/L
* Severe infection (HIV, Chronic active viral hepatitis), tests have to be conducted at screening
* Acute GvHD III-IV or extensive chronic GvHD
* The following immunosuppressive drugs (≥ 1 week of administration):

steroids ≥ 1mg/kg body weight, cytostatics (except intrathecal/ intracerebroventricular application for CNS treatment)

* Application of other experimental therapy modalities in the last 4 weeks
* Significant psychiatric disabilities, uncontrolled seizure disorders or severe peripheral neuropathy/ leukoencephalopathy
* Signs of autoimmune disease (i.e. idiopathic thrombocytopenic purpura, autoimmune hemolytic anemia)
* Subjects that do not agree to refrain from donating blood while on study drug
* Concurrent severe or uncontrolled medical disease which by assessment of the treating physician could compromise participation in the study
* Women during pregnancy and lactation
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint Part I | 49 days
  Determination of maximum tolerated dose of MOR00208 in pediatric patients
Primary endpoint Part II | 545 days
  Time until hematological relapse (> 5% leukemic blasts) or increase of MRD ≥ 2 log in bone marrow during an observation time of 545 days accounting for competing risks

SECONDARY OUTCOMES:
Pharmakokinetic of MOR00208 | 8 days
  Mean plasma concentrations of MOR00208 will be calculated and displayed graphically
Safety and toxicity of MOR00208 - Part I | 49 days
  Adverse events will be presented in line listings and also in cumulative tabulations
Treatment success | 365 days
  Rate of patients with treatment success defined as survival without newly emerging MRD or increasing MRD ≥ 2 log in bone marrow or peripheral blood or unacceptable toxicity
Overall survival | 545 days
  OS from date of first dose until end of follow up at 545 days will be analyzed using Kaplan-Meier-Methods, presenting corresponding statistical parameters and 95% confidence limits and Kaplan-Meier survival curves. Patients alive at 545 days and patients that could not be followed up until 545 days but were seen alive at the last visit will be censored.
MRD reduction | 545 days
  The amount of patients with reduction of at least 1 log at any time point compared to baseline MRD measurement between SCT and start of study treatment will be calculated and displayed graphically. Rates and 95%-confidence limits are also provided.
B cell numbers | 545 days
  Mean B cell numbers will be calculated and displayed graphically with 95%-confidence limits.
Cytotoxic lysis | 545 days
  Cytotoxic lysis will be calculated and displayed graphically.
Safety and toxicity of MOR00208 - Part II | 545 days
  Adverse events will be presented in line listings and also in cumulative tabulations

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lang, Prof., Principal Investigator — University Childrens Hospital Tübingen
Locations (11):
- Germany (11):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - University childrens Hospital, Tübingen, Baden-Wurttemberg
  - Klinik für Kinder- und Jugendmedizin, Ulm, Baden-Wurttemberg
  - Klinikum Dr. von Haunersches Kinderspital, München, Bavaria
  - Zentrum für Geburtshilfe, Kinder- und Jugendmedizin, Hamburg, Hamburg
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsmedizin Berlin, Campus Virchow Klinikum, Berlin
  - Universitätsklinikum, Essen
  - Universitätsklinikum, Klinik für Kinder- und Jugendmedizin, Frankfurt
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitäts-Kinderklinik, Würzburg

IPD SHARING:
Plan to Share IPD: No